CLINICAL TRIAL: NCT00418548
Title: A Randomized, Double-Blind, Placebo Controlled Trial Evaluating the Safety and Efficacy of Etanercept 50 mg Once Weekly Compared With 25 mg Twice Weekly in Subjects With Ankylosing Spondylitis
Brief Title: Study Comparing Etanercept 50 mg Once Weekly to 25 mg Twice Weekly in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A3-314
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2007-01-05 (Estimated); Status verified 2007-01

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The purpose of this study is to compare efficacy, pharmacokinetics, and safety of investigational formulations of etanercept administered as 50 mg once weekly with 25 mg twice weekly and placebo in patients with ankylosing spondylitis (AS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AS, as defined by Modified New York Criteria for Ankylosing Spondylitis.
* Active AS, defined by average of visual analog scale (VAS) of ≥ 30 for duration and intensity of morning stiffness and at least 2 of the following: VAS for patient global assessment ≥ 30; average of VAS for nocturnal and total pain ≥ 30; BASFI ≥ 30 (all scores on a scale of 0 to 100).

Exclusion Criteria:

* Complete ankylosis (fusion) of spine.
* Previous treatment with etanercept, antibody to Tumor Necrosis Factor α (TNFα), or other TNFα inhibitors or other biologic agents.
* Use of disease modifying antirheumatic drugs (DMARDs) other than hydroxychloroquine, sulphasalazine, and methotrexate within 4 weeks of baseline. Subjects treated with hydroxychloroquine, sulphasalazine, and methotrexate may continue these drugs during this study but doses must be held stable for 4 weeks before baseline examination and for the duration of the study.
* Receipt of multiple nonsteroidal anti-inflammatory drugs (NSAIDs) at baseline.
* Dose of NSAID changed within 2 weeks of baseline evaluation.
* Dose of prednisone >10 mg/day (or equivalent) or changed within 2 weeks of baseline evaluation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2004-06; Study Completion 2005-02

PRIMARY OUTCOMES:
The primary objective is to assess the efficacy (measured by % of subjects achieving ASAS 20 (Assessments in Ankylosing Spondylitis 20%) at week 12) and safety of etanercept 50 mg once weekly.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Baraliakos X, Szumski A, Koenig AS, Jones H. The role of C-reactive protein as a predictor of treatment response in patients with ankylosing spondylitis. Semin Arthritis Rheum. 2019 Jun;48(6):997-1004. doi: 10.1016/j.semarthrit.2018.10.019. Epub 2018 Nov 2. PMID 30473179